CLINICAL TRIAL: NCT02642185
Title: Microwave Ablation Versus Resection for Resectable Colorectal Liver Metastases
Acronym: MAVERRIC
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Freedman, Prof, Karolinska Institutet
Other Study IDs: MAVERRIC
Record Dates: First submitted 2015-10-30; First posted 2015-12-30 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neoplasm Metastasis
Keywords: microwave; ablation; resection; liver; colorectal; survival; metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ablation: Patients that are primarily treated with microwave ablation of colorectal liver metastases
  Interventions: Procedure: Microwave ablation
- Resection: Patients identified in the Swedish liver registry during the same time frame subjected to liver resection, propensity score matched to the ablation group
  Interventions: Procedure: Resection

INTERVENTIONS:
Procedure: Microwave ablation — CT-guided percutaneous ablation of 1-5, <31mm in diameter, colorectal liver metastases, performed with any generic microwave ablation system cleared for clinical use
  Groups: Ablation
Procedure: Resection — Open or laparoscopic resection of liver metastases using standard of care surgical procedures
  Groups: Resection

SUMMARY:
This study aims to prove that a strategy of first line local ablation of colorectal liver metastases with microwaves is not inferior to liver resections in terms of survival rates at three years with secondary endpoints being survival at five and ten years, interventional complication rates, length of stay, ablation precision measurements, need for further interventions and health-economic analysis.

A cohort of 100 patients treated with CT guided microwave ablation of 1-5 metastases <31mm in size will be followed and compared with propensity scored matched controls from the Swedish liver surgery registry - Sweliv.

The study is a multi-institutional effort by the Hepato Pancreatico Biliary (HPB) units in Stockholm Sweden, Bern Switzerland and Groningen in the Netherlands.

DETAILED DESCRIPTION:
BACKGROUND

Surgery Surgical resection of operable colorectal liver metastases is the current gold standard. With advancement in surgical techniques and technology the 3-year survival rate for this group of patients is now in the range of 60% [1] where the survival without resection is virtually non-existent. Palliative chemotherapy can prolong survival for 12-24 months, but very rarely much more than this [2].

Operability is decided by the general health condition of the patient, the global liver function and tumour associated factors like the number, size and distribution of the liver metastases.

It is uncommon to disqualify surgery because of the general health of the patient, but is sometimes a reality with advanced age and severe comorbidities.

The combination of size, number and distribution of liver metastases determines the extent of the resection and thereby the size of the liver that will remain after surgery. This is a critical factor as postoperative liver failure is often fatal. With an otherwise healthy liver, approximately 75% of the parenchyma can be resected and the remaining 25% will within a year has regenerated so that the total liver volume is around 80-90% of the original liver [3].

This regenerative capacity is used to make complex resections in stages, there by manipulating an initially small liver remnant to a sufficient size for survival.

Liver surgery, however, comes with a price. For small local resections and laparoscopic minor hepatectomies the morbidity of surgery is 20-30% with a quarter being serious. For major and complex procedures the morbidity is 40-50% with the same proportion of serious complications requiring further surgical intervention or death [4]. With advanced patient support and state of the art surgical technique, the mortality following surgery is small, typically in the range of 1-2%.

The patients spend 5-14 days in hospital and are incapacitated for a month or two after open surgery, significantly less after laparoscopic surgery where the patient usually can return home after 2-7 days in hospital and with an early return to normal physical activities within two weeks.

Another factor to take into account is the frequency of liver recurrences. After resection, 50-80% of the patients will get new liver metastases [5]. With previous major resections the choice of following surgical strategies gets more limited.

Ablations Local ablation techniques have evolved from local injection of cytotoxic agents like ethanol and acetic acid to thermal ablations with freezing of the tissue or heating with radiofrequency energy, laser beams or microwave energy. Ablations can also be done by destroying cell membranes with electricity in short intense bursts, the irreversible electroporation technique, causing localised cell death with very little heat thereby preserving collagen structures and other surrounding proteins, which will result in patent vessels, bile-ducts and nerve sheaths [6].

The ablative procedures have two critical points; the correct localization of the energy and the correct amount of energy. Ablation in the wrong place will decrease the efficacy as will an incorrect size of the ablation.

Targeting of lesions has improved with computer assisted targeting and fusion of radiological modalities so that as much information as possible can be used in the placement of the energy source. Percutaneous ultrasound targeting has until recently been the most common means of placing ablation devices in liver lesions. Local recurrence rates of 20-30% are typically reported with this approach. With more recent fused and computer assisted techniques the local recurrence rate is often stated to be around 5-10% [7].

The main limitation with ablative techniques is the size of the lesions. Many studies have shown a good result with lesion less than 30mm in diameter and increasing recurrence rates with larger lesions. A single ablation can usually only be up to 40-50mm in diameter. Larger lesions can be treated with multiple applications but the geometries of ovoid ablations in irregular tumours makes complete ablations difficult.

Destroying lesions with ablative techniques spares liver parenchyma and allows for treating patients that are not resectable in situations with multiple lesions engaging all or most of the liver segments. This approach has greatly increased the survival in this group of patients. Sparing unaffected liver parenchyma also increases the flexibility when there are liver recurrences of metastatic disease. This happens in up to 50 percent of patients after local resections and ablations and in a third of patients after major hepatectomies and with a focused ablative approach more functioning liver parenchyma can be saved and the options for treatment of recurrences are wider.

Lesions can be targeted with a percutaneous approach using ultrasound fused with magnetic resonance imaging or computer tomography, or in the CT with guidance techniques, or laparoscopically if needed. Very rarely an open approach is needed.

This means that patients usually goes home the same day or the day after treatment and has returned to normal physical activities within a week.

Morbidity is in the area of 10% with a fourth being serious complications requiring some kind of intervention. Mortality is typically very low and under 1%.

Local thermal ablations have been shown to be equal to resections in the treatment in hepatocellular carcinoma when lesions are less than 30mm in size. These data come from retrospective analyses of single centre experiences and are as such of low scientific grade of evidence [8,9].

Study design considerations There has not been any well-powered randomized study comparing an ablative strategy with a resective. Doing a non-inferiority randomized study with sufficient power would need up to a thousand patients in each group, thus making this study virtually impossible to conduct. A way to come around this is to use propensity score techniques to compare cases with controls. The investigators have well documented controls in the swedish liver registry allowing for propensity score matching of the data.

With this design only 100 patients will have to be treated, as has been computed with a power calculation with survival curves after resective treatment with colorectal liver metastases. Data was extracted from "Livermet survey", an on-line prospective database with more than 25000 hepatectomies for colorectal cancer in 69 countries. Data for a first resection of a single metastasis smaller than 30mm (best case scenario) was extracted and survival curves computed. With a non-inferiority assumption, with a power of 90% and the non-inferiority limit being not worse than 5% reduction in 3-year survival, a sample size of 100 was computed, see figure below.

CLINICAL AND ECONOMICAL CONSEQUENCES If the study thesis holds there would be a great impact on the treatment of colorectal liver metastases where approximately half could be treated with a minimal invasive and low-complication ablation strategy, greatly reducing patient morbidity and increasing possibilities for further treatment modalities in case of tumour recurrences in the liver. With much shorter hospital stay and sick-leave there is a great potential for big savings in health-related costs for health service providers.

From Engstrand et al. In manuscript. This shows the distribution of 272 liver metastases from colorectal cancer among a population based cohort of 1032 patients that were diagnosed with that primary in the greater Stockholm area in 2008. Approximately half of all patients eligible for resection could potentially be treated with ablation.

STUDY DESIGN European multicentre prospective cohort study with propensity score matching for number or tumours, age, gender and response to chemotherapy (no chemo - response/stable disease - progression).

Patients with colorectal liver metastases are evaluated at a weekly liver multidisciplinary conference and a treatment strategy is decided. In this decision process patients that are resectable and have tumours of 30mm or less and not more than 5 in number, and deemed as both ablatable and resectable, will be offered treatment with an ablative strategy using state of the art targeting and microwave ablation devices. During the study inclusion phase, which can be sequential or with specific weeks during the year (one in two/three/four/five depending on local considerations), all patients that fulfill the inclusion criteria must be entered into the database. All ablations will be done with computer assisted CT targeting (Cascination AG, Bern, Ch) allowing for precise image documentation and evaluation of tumour, ablation device placement and resulting ablation zones. Repeat ablation is allowed and a new multidisciplinary team conference (MDT) discussion is mandated with loss of disease control.

Patient characteristics and procedure related parameters will be recorded and outcome measured as overall survival at three years using survival analysis. Secondary outcomes will be tumour state (disease free interval), complications, local recurrence rates, accuracy in placement of ablative device, analyses of ablation volumes, length of stay and further need of treatment with ablations or resections.

Treatment with chemotherapy will be as decided at the MDT and with the same protocol that is used with neoadjuvant or adjuvant treatment with surgical resection.

Patients will give their informed consent before entering the study.

Patient data will be stored in a secure password-protected server with Red-cap software belonging to Karolinska Institutet at Danderyd Hospital. Procedural data will be stored together with image series downloaded directly from the ablation aiming device to Artorg Centre at the University of Bern, responsible for volumetric and precisional data analyses in the study.

Patient recruitment will primarily be from the greater Stockholm area. All treatment of swedish patients will be at Danderyd Hospital, Stockholm Sweden.

A second centre will be at Inselspital in Bern, Switzerland, and a third in Groningen in the Netherlands.

With an optimal inclusion rate the study will have recruited the necessary patients within one year.

TIME FRAME September 1: finalization of protocol and submission to ethics board November 2015: Start inclusion November 2017?: Inclusion complete 2018: Publication of intervention specific data like workflow, precision and ablation volumes.

2020: Three year follow-up finished and files closed for main study 2021: Publication of results 2023: Evaluation and publication of 5-year survival data 2028: Evaluation and publication of 10-year survival data. Database finally closed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1-5 colorectal liver metastases
* No metastases larger than 30 mm in diameter
* All lesions amenable to CT-guided percutaneous microwave ablation
* Patient also resectable
* Patients so evaluated at the multidisciplinary tumor board meeting

Exclusion Criteria:

* Kidney failure excluding the use of iv contrast medium
* Lack of informed consent
* Logistic reasons where patient does not live in the region of the treatment centre

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European multicentre prospective cohort study with propensity score matching for number or tumours, age, gender and response to chemotherapy (no chemo - response/stable disease - progression).
  Patients with colorectal liver metastases are evaluated at a weekly liver multidisciplinary conference and a treatment strategy is decided. In this decision process patients that are resectable and have tumours of 30mm or less and not more than 5 in number, and deemed as both ablatable and resectable, will be offered treatment with an ablative strategy using state of the art targeting and microwave ablation devices.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Overall survival | 10 years
Complications to treatment | 1 year
Disease free survival | 3 years
Overall cost of treatment as measured in euros | 3 years
  The aggregated health provider's costs for all liver specific treatments including index surgery and hospital costs, costs for further liver specific interventions.
Local recurrence rates | 3 years
Accuracy of placement of ablative device measured as mm from needle target location | intraoperative
Analysis of ablation volumes measured as length and radius of ovoid ablation zone. | 1-28 days post intervention
Need for further liver specific treatment as assessed by number of sessions with ablation or resections | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Freedman, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- University Medical Centre, Groningen, Netherlands
- Karolinska Institutet, Dept of Surgery at Danderyd Hospital, Stockholm, Sweden
- Pascale Tinguely, Bern, Switzerland

REFERENCES:
- [Background] www.livermetsurvey.com, annual statistics june 2014.
- [Background] Costi R, Leonardi F, Zanoni D, Violi V, Roncoroni L. Palliative care and end-stage colorectal cancer management: the surgeon meets the oncologist. World J Gastroenterol. 2014 Jun 28;20(24):7602-21. doi: 10.3748/wjg.v20.i24.7602. PMID 24976699
- [Background] Pomfret EA, Pomposelli JJ, Gordon FD, Erbay N, Lyn Price L, Lewis WD, Jenkins RL. Liver regeneration and surgical outcome in donors of right-lobe liver grafts. Transplantation. 2003 Jul 15;76(1):5-10. doi: 10.1097/01.TP.0000079064.08263.8E. PMID 12865779
- [Background] Dokmak S, Fteriche FS, Borscheid R, Cauchy F, Farges O, Belghiti J. 2012 Liver resections in the 21st century: we are far from zero mortality. HPB (Oxford). 2013 Nov;15(11):908-15. doi: 10.1111/hpb.12069. Epub 2013 Mar 6. PMID 23461811
- [Background] Jones NB, McNally ME, Malhotra L, Abdel-Misih S, Martin EW, Bloomston M, Schmidt CR. Repeat hepatectomy for metastatic colorectal cancer is safe but marginally effective. Ann Surg Oncol. 2012 Jul;19(7):2224-9. doi: 10.1245/s10434-011-2179-0. Epub 2011 Dec 30. PMID 22207046
- [Background] Nosher JL, Ahmed I, Patel AN, Gendel V, Murillo PG, Moss R, Jabbour SK. Non-operative therapies for colorectal liver metastases. J Gastrointest Oncol. 2015 Apr;6(2):224-40. doi: 10.3978/j.issn.2078-6891.2014.065. PMID 25830041
- [Background] Pathak S, Jones R, Tang JM, Parmar C, Fenwick S, Malik H, Poston G. Ablative therapies for colorectal liver metastases: a systematic review. Colorectal Dis. 2011 Sep;13(9):e252-65. doi: 10.1111/j.1463-1318.2011.02695.x. PMID 21689362
- [Background] Osaki Y, Nishikawa H. Treatment for hepatocellular carcinoma in Japan over the last three decades: Our experience and published work review. Hepatol Res. 2015 Jan;45(1):59-74. doi: 10.1111/hepr.12378. Epub 2014 Jul 18. PMID 24965914
- [Background] Park EK, Kim HJ, Kim CY, Hur YH, Koh YS, Kim JC, Kim HJ, Kim JW, Cho CK. A comparison between surgical resection and radiofrequency ablation in the treatment of hepatocellular carcinoma. Ann Surg Treat Res. 2014 Aug;87(2):72-80. doi: 10.4174/astr.2014.87.2.72. Epub 2014 Jul 29. PMID 25114886